CLINICAL TRIAL: NCT03432650
Title: Evaluation of Anterior Quadratus Lumborum Block for Postoperative Analgesia in Hip Arthroscopy: A Double-Blinded Randomized Controlled Trial
Brief Title: Evaluation of Anterior Quadratus Lumborum Block for Postoperative Analgesia in Hip Arthroscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-0647
Record Dates: First submitted 2018-01-25; First posted 2018-02-14 (Actual); Results first posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-07

CONDITIONS: Hip Disease
MeSH Terms: interventions — Bupivacaine; Dexamethasone; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QLB Block + Standard of Care (Experimental): Patients will receive either a spinal (4cc Mepivacaine) or combined spinal epidural anesthetic (dose up 50 5 cc 2% lidocaine) with IV sedation. Intraoperative anti-emetics will consist of IV ondansetron and IV dexamethasone. Intra-operative analgesics will be IV fentanyl, IV acetaminophen, IV ketorolac, and IV ketamine. No Block will be given.
  Patients will receive a single shot anterior QLB (30cc 0.5% Bupivacaine with 2mg preservative free dexamethasone).
  Interventions: Drug: Bupivacaine + dexamethasone; Device: Ultrasound
- Standard of Care (No Intervention): Patients will receive either a spinal (4cc Mepivacaine) or combined spinal epidural anesthetic (dose up 50 5 cc 2% lidocaine) with IV sedation. Intraoperative anti-emetics will consist of IV ondansetron and IV dexamethasone. Intra-operative analgesics will be IV fentanyl, IV acetaminophen, IV ketorolac, and IV ketamine. No Block will be given.

INTERVENTIONS:
Drug: Bupivacaine + dexamethasone — Anesthetic that will help treat pain and sensation after hip arthroscopy
  Arms: QLB Block + Standard of Care
Device: Ultrasound — Ultrasound will help guide the anesthesiologist in performing the nerve block
  Arms: QLB Block + Standard of Care

SUMMARY:
Hip arthroscopy is performed frequently and the postoperative course often involves moderate to severe pain. There remains no definitive perioperative pain regimen that has been proven to be effective and safe for this ambulatory procedure. Some institutions perform peripheral nerve blocks either preoperatively or postoperatively as a rescue block. All of these PNBs lead to quadriceps weakness which may impede earlier mobilization and physical therapy. While some case reports exist, there have not been any studies evaluating the QLB for hip arthroscopy patients. As previously mentioned, the technique is easy to perform, well-tolerated by patients, and avoids side effects such as hypotension, urinary retention, or the quadriceps weakness associated with lumbar plexus blockade.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for hip arthroscopy
* Ability to follow study protocol
* English Speaking

Exclusion Criteria:

* Hepatic or renal insufficiency
* Younger than 18 years old and older than 80
* Allergy or intolerance to one of the study medications
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (daily opioids use for longer than 3 months)
* Patients contraindicated to undergo a spinal anesthetic
* Non English Speakers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Haskins, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital of Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- QLB Block + Standard of Care: Patients will receive either a spinal (4cc Mepivacaine) or combined spinal epidural anesthetic (dose up 50 5 cc 2% lidocaine) with IV sedation. Intraoperative anti-emetics will consist of IV ondansetron and IV dexamethasone. Intra-operative analgesics will be IV fentanyl, IV acetaminophen, IV ketorolac, and IV ketamine. No Block will be given.
  Patients will receive a single shot anterior QLB (30cc 0.5% Bupivacaine with 2mg preservative free dexamethasone).
  Bupivacaine + dexamethasone: Anesthetic that will help treat pain and sensation after hip arthroscopy
  Ultrasound: Ultrasound will help guide the anesthesiologist in performing the nerve block
Period: Overall Study
Arm/Group | QLB Block + Standard of Care | Standard of Care
Started | 48 | 48
Completed | 48 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QLB Block + Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (13) | 36 (12) | 36 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 22 | 24 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 26 (5.7) | 24.9 (3.8) | 25 (4.9)
Short Form-8 Health Questionnaire [Mean (Standard Deviation); unit: units on a scale] — This questionnaire consists of 8 questions. The score for each question is 1-5. a lower score is a better outcome. maximum score is 40, minimum score is 8. scores are reported the total for all 8 questions combined.
  units on a scale | 16 (4) | 17 (6) | 16.4 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Numerical Pain Rating System (NRS) Pain Scores
Description: Pain scores at rest and with movement will be through 24 hours after surgery. Score scale is from 0-10. 0 means no pain, 10 means worst pain. A lower score is a better outcome.
Time Frame: 30min after Post Anesthesia Care Unite (PACU) arrival
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
score on a scale
  NRS at Rest | 3.3 (3.4) | 4.4 (3.3)
  NRS with Movement | 4.5 (4) | 4.7 (3.6)

2. Primary Outcome: Numerical Pain Rating System (NRS) Pain Scores
Description: as for outcome 1
Time Frame: 1 hour after Post Anesthesia Care Unite (PACU) arrival
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
score on a scale
  NRS at Rest | 3.7 (3.2) | 4.6 (3.7)
  NRS with Movement | 4.1 (3.2) | 5.2 (2.9)

3. Primary Outcome: Numerical Pain Rating System (NRS) Pain Scores
Description: as for outcome 1
Time Frame: 2 hours after Post Anesthesia Care Unite (PACU) arrival
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
score on a scale
  NRS at Rest | 4.1 (2.1) | 4.6 (2.4)
  NRS with Movement | 4.5 (2.3) | 4.8 (2.5)

4. Primary Outcome: Numerical Pain Rating System (NRS) Pain Scores
Description: as for outcome 1
Time Frame: 3 hours after Post Anesthesia Care Unite (PACU) arrival
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
score on a scale
  NRS at Rest | 4.1 (2.3) | 4.6 (2.2)
  NRS with Movement | 4.6 (2.3) | 4.8 (2.4)

5. Primary Outcome: Numerical Pain Rating System (NRS) Pain Scores
Description: as for outcome 1
Time Frame: 24 hours after Post Anesthesia Care Unite (PACU) arrival
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
score on a scale
  NRS at Rest | 3.3 (2.5) | 3.8 (2.1)
  NRS with Movement | 5.7 (2.6) | 5.7 (2.3)

6. Secondary Outcome: Opioid Use
Description: Amount of opioids taken after surgery
Time Frame: After Surgery to Post Operative Day 1
Measure: Median (Inter-Quartile Range); unit: oral morphine equivalent units (mg)
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
oral morphine equivalent units (mg) | 75 [41 to 90] | 68 [45 to 75]

7. Secondary Outcome: Number of Patients With Presence of IAFE (Intraabdominal Fluid Extravasation) Following Surgery
Time Frame: Immediately post-op in OR
Measure: Count of Participants; unit: Participants
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
Participants | 9 | 11

8. Secondary Outcome: Number of Patients With Nausea/Vomiting
Time Frame: Up to Post Op Day 1
Population: some patients did not answer survey questions
Measure: Count of Participants; unit: Participants
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
Participants
  Nausea PACU: number analyzed (Participants) | 48 | 45
  Nausea PACU | 12 | 7
  Nausea POD1 (24hr): number analyzed (Participants) | 45 | 45
  Nausea POD1 (24hr) | 21 | 19
  Vomiting PACU: number analyzed (Participants) | 48 | 45
  Vomiting PACU | 0 | 1
  Vomiting POD1 (24hr): number analyzed (Participants) | 45 | 45
  Vomiting POD1 (24hr) | 2 | 3

9. Secondary Outcome: Antiemetic Use
Time Frame: Up to Post Op Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
Participants | 18 | 12

10. Secondary Outcome: Number of Participants With Hospital Admission
Time Frame: Up to Post Op Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
Participants | 11 | 9

11. Secondary Outcome: Patient Satisfaction With Post Op Pain Control
Description: Scale of 0-10; 0 being extremely dissatisfied and 10 being extremely satisfied
Time Frame: Up to Post Op Day 1
Population: some patients did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
score on a scale
  PACU: number analyzed (Participants) | 47 | 45
  PACU | 8 (2) | 9 (2)
  POD1: number analyzed (Participants) | 48 | 45
  POD1 | 8 (2) | 9 (2)

12. Secondary Outcome: Patient Score on Quality of Recovery-40 (QoR40) Inventory.
Description: Validated QoR40 survey score. Survey questions are added up to provide a final score. Higher score is reflective of a better outcome. Minimum score is 40, maximum score is 200.
Time Frame: Up to Post Op Day 1
Population: Some patients did not answer questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 46 | 46
score on a scale
  PACU | 104.9 (7) | 107.5 (7.1)
  POD1: number analyzed (Participants) | 45 | 45
  POD1 | 105.6 (7.4) | 105 (7.3)

13. Secondary Outcome: Change in Quadriceps Motor Strength on Surgical Side
Description: Change in Quadriceps Motor Strength from Pre-Op Baseline Quadriceps Strength
Time Frame: Up to Post Op Day 1
Population: some patients were lost to follow up
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 27 | 30
kg | -4.4 (3.3) | -3.5 (2.4)

14. Secondary Outcome: Urinary Retention
Description: Incidence of Urinary Retention in recovery
Time Frame: Up to Post Op Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
Participants | 1 | 0

15. Secondary Outcome: Incidence of Hypotension
Time Frame: Up to Post Op Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | QLB Block + Standard of Care | Standard of Care
Number analyzed (Participants) | 48 | 48
Participants | 16 | 19

ADVERSE EVENTS:
Time Frame: 6 months following surgery
Arm/Group | QLB Block + Standard of Care | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT03432650/Prot_SAP_000.pdf